CLINICAL TRIAL: NCT03507010
Title: Ledderhose Disease: Radiotherapy or Not? A Randomised, Multicentre, Prospective, Double Blind Phase III Trial Investigating the Effect of Radiotherapy on Patients With Ledderhose Disease
Brief Title: Ledderhose Disease: Radiotherapy or Not?
Acronym: LedRad
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Catharina Ziekenhuis Eindhoven (Other); Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RT2015-03
Record Dates: First submitted 2018-02-27; First posted 2018-04-24 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Ledderhose Disease
Keywords: Radiotherapy; Pain
MeSH Terms: conditions — Fibromatosis, Plantar; Pain | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy (Experimental): Patients assigned to the Radiotherapy group are treated with electrons and will receive a total dose of 30 Gy.
  Interventions: Radiation: Radiotherapy
- Sham Radiotherapy (Placebo Comparator): Patients assigned to the sham-radiotherapy group will not actually receive radiation. For these patients the radiation is simulated.
  Interventions: Other: Sham Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Patients randomized to the Radiotherapy arm will be treated with electrons and receive a total dose of 30 Gy (two separate courses of five daily fractions of 3.0 Gy each).
  Arms: Radiotherapy
Other: Sham Radiotherapy — Patients randomized to the sham-radiotherapy will not be treated and the radiotherapy treatment will only be simulated.
  Arms: Sham Radiotherapy

SUMMARY:
The aim of the LedRad trial is to determine the efficacy and durability of radiotherapy as treatment for patients with Ledderhose disease and to compare this to the natural course of Ledderhose disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful Ledderhose disease. The pain score measured with the VAS score and is at least 2 on the 11-point scale (0 = no pain to 10 = worst imaginable pain).
* Age ≥ 18 years
* WHO performance status 0, 1 or 2 (Appendix, section 18)
* Before patient randomisation, written informed consent must be given according to ICH/GCP, and WMO requirements.
* Controlling the Dutch language (speaking and reading).
* Able and willing to complete quality of life questionnaires in Dutch
* Must be accessible for treatment follow-up

Exclusion Criteria:

* Surgical intervention before for Ledderhose disease
* Previous radiation treatment for Ledderhose disease
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Not able to lay prone for at least fifteen minutes
* Females who are pregnant at entry or who want to become pregnant within six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2029-03-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale | 12 months
  Determine pain with the Numeric Rating Scale

SECONDARY OUTCOMES:
Numeric Rating Scale | 6 and 18 months
  Determine pain with the Numeric Rating Scale
Size of ledderhose nodules | 12 months
  Determine the effect of radiotherapy on size of Ledderhose nodules with MRI and Ultrasound
Walking distance | 6, 12 and 18 months
  Determine the effect of radiotherapy on walking distance with the 10 meter straight line walk test
Walking motion | 12 months
  Determine the effect of radiotherapy on walking motion with the PEDAR-X® in shoe pressure measurement system
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 18 months
  Assess the safety and toxicity of radiotherapy on this population by recording the toxicity of radiotherapy during the course of radiotherapy and thereafter measured by CT-CAE 4.0.
Quality of life (1) | 6, 12 and 18 months
  Assess the impact on quality of life of radiotherapy as treatment for this study population with RAND-36 item Health Survey questionnaire
Quality of life (2) | 6, 12 and 18 months
  Assess the impact on quality of life of radiotherapy as treatment for this study population with the brief pain inventory questionnaire
Quality of life (3) | 6, 12 and 18 months
  Assess the impact on quality of life of radiotherapy as treatment for this study population with the EURO-Qol-5D questionnaire
Cost-effectiveness analysis (CEA) | 6, 12 and 18 months
  The economic evaluation will be performed from a societal perspective, incorporating cost of travel to the hospital and cost of absence from work as well as direct medical cost of radiotherapy (cost of irradiation and outpatient visits). Questionnaires will be used to collect data regarding health care consumption, travel and time costs, and productivity loss at study entry and at 6-month intervals thereafter. In addition to the pain scores, quality of life will be assessed at 6-month intervals using the Rand-36 questionnaire. The utilities based on the results of the questionnaire will be used in a cost-utility analysis, calculating the ratio of incremental costs versus incremental quality-adjusted life-years (QALY).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No